CLINICAL TRIAL: NCT03562065
Title: Treatment of Refractory Systemic Lupus Erythematosus by Injection of Allogeneic Mesenchymal Stem Cells Derived From the Umbilical Cord
Brief Title: Treatment of Refractory Systemic Lupus Erythematosus by Allogeneic Mesenchymal Stem Cells Derived From the Umbilical Cord
Acronym: MSC-SLE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150302
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Lupus Erythematosus; Stem Cell Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mesenchymal stem cells (Experimental): Phase I-II, Allogeneic Umbilical Cord derived-MSCs injected by slow intravenous infusion according to the weight of the recipient and patient groups in the study, at doses of:
  * 1.10^6 CSM / kg
  * 2.10^6 CSM / kg
  * 4.10^6 CSM / kg 1 injection during 30min to 1h by Intravenous infusion
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — Allogeneic Umbilical Cord derived-MSCs injected by slow intravenous infusion according to the weight of the recipient and patient groups in the study, at doses of:
  * 1.10^6 CSM / kg
  * 2.10^6 CSM / kg
  * 4.10^6 CSM / kg 1 injection during 30min to 1h by Intravenous infusion

SUMMARY:
Systemic lupus erythematosus (SLE) is a rare (prevalence: 40- 50/100 000 persons) heterogeneous auto-immune and auto-inflammatory disease (AD), affecting both sexes and all races, with a peak incidence / prevalence among black people and a predilection for women in the 3rd-4th decade of life. SLE is characterized by successive periods of flares and remission, which may all vary in duration and quality. Prognosis of severe forms of SLE, which affect lung, heart or brain in addition to renal involvement, has improved, but still evolution remains pejorative in a subset of patients whose 10 years mortality remains 10-15%, even in tertiary referral centers. For 20 years, no new prospective clinical trial in the course of SLE has demonstrated its effectiveness. New biological therapies have not yet made the long awaited breakthrough in the treatment of severe SLE and only anti-Blys monoclonal antibody has gained indication in moderately active SLE. In addition, serious adverse side effects (progressive multifocal leukoencephalopathy) observed with several biologics in AD patients has dampened their expected benefits. For SLE subjects resistant to 1er or 2nd line conventional treatment, there is a need to develop more effective therapies with fewer long term side effects, based on new immunomodulatory and immunosuppressive strategies.

According to their in vitro immunomodulatory properties and ability to induce tissue repair mechanisms, mesenchymal stem cells (MSC) have been proposed as a new therapy for several AD, including SLE. The use of allogeneic umbilical cord-derived MSC is based on experimental and human clinical data, particularly produced by Nanjing team (Pr Sun) in China. It is also logical to select SLE patients with the same severity criteria as those used worldwide to validate the efficacy of anti-Blys therapies. Similarly, the analysis of the expected results should take into account criteria similar or comparable to those used for the pivotal clinical trials. This trial is a unique opportunity to set up collaboration between Saint-Louis APHP, clinical expert center for cell therapy in AD, and University College London for cell manufacturing.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 70 years.
* Diagnosis of Systemic Lupus Erythematosus (SLE) according to the ACR criteria with positive antinuclear antibodies.
* Subjects with sustained disease activity defined by a SELENA- SLEDAI SLE activity index ≥ 6 at baseline,
* Inefficacy or adverse effects necessitating discontinuation of first and second line therapies of SLE including:

  a. Prednisone orally ≥ 6 mg / day (or equivalent) for at least 28 days. b. At least one or more of the following immunosuppressive therapies for 3 months in total: i- Cyclophosphamide, iv bolus ≥500 mg / month for 3 months minimum ii- Mycophenolate mofetil, orally or equivalent at a dose> 2000 mg / day for at least 90 days iii- Azathioprine orally at a dose> 2 mg / kg / day for at least 90 days; iv- Methotrexate orally or parenterally, at doses > 20mg / week for at least 90 days; v- Leflunomide orally, at a dose of> 10-mg / day for at least 90 days; vi- Rituximab (anti-CD20) intravenous bolus 375 mg / m2, once a week for four weeks or total dose of 1 g twice a day for two weeks vii- Cyclosporine orally, at a dose of 2.5-5 mg / kg / day, for at least 90 days; viii- Belimumab intravenously at monthly bolus of 10 mg / kg infusion), for at least 3 months.
* Patient who received treatment of SLE at stable doses for a minimum of 30 days prior to eligibility, including one of the following treatments: prednisone (or equivalent) alone or combined with antimalarial treatment, an anti-inflammatory steroidal and / or an immunosuppressant.
* Negative pregnancy test for women of childbearing age.
* For men and women : Using effective contraceptive methods during treatment and within 3 months after the end of treatment for men with her partner of childbearing age
* Signed Informed Consent.
* Affiliation to social security.

Exclusion Criteria:

1- Pregnancy, breastfeeding or lack of appropriate contraception during study duration

* Presence of:

  1. Renal failure: calculated creatinine clearance of <30 ml / min
  2. Cardiac failure: clinical signs of congestive heart failure; left ventricular ejection fraction <40% on echocardiography; uncontrolled ventricular arrhythmia;
  3. Hepatitis defined by abnormal levels of transaminases (AST, ALT> 2 x normal) not related to disease activity.
  4. Respiratory disease: mean PAP> 50 mmHg (echocardiography), respiratory failure defined by a resting blood pressure of oxygen at PaO 2 < 70 mmHg and / or PaCO2 > 50 mmHg without oxygen
* Severe psychiatric disorders, including severe psychosis related to SLE, which would prevent to give informed consent or to undergo the procedure.
* Active neoplasia or concomitant myelodysplasia, except for basal cell carcinoma or squamous cell carcinoma or in situ cervix carcinoma.
* Bone marrow failure defined by neutropenia <0.5.109/L, thrombocytopenia <30. 109 / L, anemia < 8 g / dL, lymphopenia CD4 + <200 x 106 / L caused by another disease than SLE.
* Acute or chronic uncontrolled infection: HIV 1/2, HTLV-1/2, Hepatitis B (HBsAg surface antigen), Hepatitis C with positive PCR
* Patient having received belimumab within 2 months of belimumab within 2 months of Baseline, or having received rituximab or other B cell depleting biologic therapy within 6 months of Baseline
* Current substance abuse or recent (within 60 days) history of substance abuse
* Patient in periods of exclusion from the national roster of researchers
* Patient with Linguistic or psychological incapacity to sign informed consent
* Patient already included in another study at the same time.
* Poor patient compliance.
* Patient under legal protection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity of allogeneic MSC injection according to CTCAE | 10 days
  Immediate tolerance as assessed after the first allogeneic MSC injection, according to standards CTCAE side effects. An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3.

SECONDARY OUTCOMES:
Toxicity of allogeneic MSC injection according to CTCAE Month 1 | 1 month
  Tolerance according to side effects defined by CTCAE standards (Miller Results of cancer treatment Cancer 1981; 47 (1): 207 - 214). Treatment-related toxicity will be analyzed according to the international World Health Organization (WHO) (maximum degree of toxic attacks by the body). An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3.
Toxicity of allogeneic MSC injection according to CTCAE Month 3 | 3 months
  Tolerance according to side effects defined by CTCAE standards (Miller Results of cancer treatment Cancer 1981; 47 (1): 207 - 214). Treatment-related toxicity will be analyzed according to the international World Health Organization (WHO) (maximum degree of toxic attacks by the body). An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3.
Toxicity of allogeneic MSC injection according to CTCAE Month 6 | 6 months
  Tolerance according to side effects defined by CTCAE standards (Miller Results of cancer treatment Cancer 1981; 47 (1): 207 - 214). Treatment-related toxicity will be analyzed according to the international World Health Organization (WHO) (maximum degree of toxic attacks by the body). An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3.
Toxicity of allogeneic MSC injection according to CTCAE Month 12 | 12 months
  Tolerance according to side effects defined by CTCAE standards (Miller Results of cancer treatment Cancer 1981; 47 (1): 207 - 214). Treatment-related toxicity will be analyzed according to the international World Health Organization (WHO) (maximum degree of toxic attacks by the body). An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3.
Proportion of subjects with Clinical Response Month 3 | 3 months
  Proportion of subjects with Major Clinical Response (MCR) and the proportion of subjects with Partial Response Clinic (PCR)
Proportion of subjects with Clinical Response Month 6 | 6 months
  Proportion of subjects with Major Clinical Response (MCR) and the proportion of subjects with Partial Response Clinic (PCR)
Proportion of subjects with Clinical Response Month 9 | 9 months
  Proportion of subjects with Major Clinical Response (MCR) and the proportion of subjects with Partial Response Clinic (PCR)
Proportion of subjects with Clinical Response Month 12 | 12 months
  Proportion of subjects with Major Clinical Response (MCR) and the proportion of subjects with Partial Response Clinic (PCR)
Disease activity measured by the BILAG index Month 3 | 3 months
  Disease activity measured by the British Isles Lupus Assessment Group (BILAG) index (min=0 to max=72). The higher value is the higher is the disease activity.
Disease activity measured by SELENA-SLEDAI Month 3 | 3 months
  Disease activity measured by the Safety of Estrogens in Lupus National Assessment study (SELENA) of the Systemic lupus erythematosus disease activity index (SLEDAI) (min=0 to max=105). The higher value is the higher is the disease activity.
Disease activity measured by SELENA-SLEDAI Month 6 | 6 months
  Disease activity measured by the Safety of Estrogens in Lupus National Assessment study (SELENA) of the Systemic lupus erythematosus disease activity index (SLEDAI) (min=0 to max=105). The higher value is the higher is the disease activity.
Disease activity measured by the BILAG index Month 6 | 6 months
  Disease activity measured by the British Isles Lupus Assessment Group (BILAG) index (min=0 to max=72). The higher value is the higher is the disease activity.
Disease activity measured by the BILAG index Month 9 | 9 months
  Disease activity measured by the British Isles Lupus Assessment Group (BILAG) index (min=0 to max=72). The higher value is the higher is the disease activity.
Disease activity measured by SELENA-SLEDAI Month 9 | 9 months
  Disease activity measured by the Safety of Estrogens in Lupus National Assessment study (SELENA) of the Systemic lupus erythematosus disease activity index (SLEDAI) (min=0 to max=105). The higher value is the higher is the disease activity.
Disease activity measured by the BILAG index Month 12 | 12 months
  Disease activity measured by the British Isles Lupus Assessment Group (BILAG) index (min=0 to max=72). The higher value is the higher is the disease activity.
Disease activity measured by SELENA-SLEDAI Month 12 | 12 months
  Disease activity measured by the Safety of Estrogens in Lupus National Assessment study (SELENA) of the Systemic lupus erythematosus disease activity index (SLEDAI) (min=0 to max=105). The higher value is the higher is the disease activity.
SRI Month 3 | 3 months
  SRI (Systematic lupus erythematosus Responder Index) response rate during follow-up. A SRI response is defined as a binary outcome equal to 1 if all following conditions are validated:
  * 4 points reduction of SELENA SLEDAI-score
  * no new BILAG A score for an organ
  * no more than one new BILAG B score
  * no worsening in the overall evaluation of the physician as compared to inclusion values
SRI Month 6 | 6 months
  SRI (Systematic lupus erythematosus Responder Index) response rate during follow-up. A SRI response is defined as a binary outcome equal to 1 if all following conditions are validated:
  * 4 points reduction of SELENA SLEDAI-score
  * no new BILAG A score for an organ
  * no more than one new BILAG B score
  * no worsening in the overall evaluation of the physician as compared to inclusion values
SRI Month 9 | 9 months
  SRI (Systematic lupus erythematosus Responder Index) response rate during follow-up. A SRI response is defined as a binary outcome equal to 1 if all following conditions are validated:
  * 4 points reduction of SELENA SLEDAI-score
  * no new BILAG A score for an organ
  * no more than one new BILAG B score
  * no worsening in the overall evaluation of the physician as compared to inclusion values
SRI Month 12 | 12 months
  SRI (Systematic lupus erythematosus Responder Index) response rate during follow-up. A SRI response is defined as a binary outcome equal to 1 if all following conditions are validated:
  * 4 points reduction of SELENA SLEDAI-score
  * no new BILAG A score for an organ
  * no more than one new BILAG B score
  * no worsening in the overall evaluation of the physician as compared to inclusion values
comorbidities Month 3 | 3 months
  Presence of comorbidities
comorbidities Month 6 | 6 months
  Presence of comorbidities
comorbidities Month 9 | 9 months
  Presence of comorbidities
comorbidities Month 12 | 12 months
  Presence of comorbidities
Quality of life Month SF-36 Month 3 | 3 months
  Quality of life assessed by the Short Form 36 version 2 (SF-36v2). The SF-36v2 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life EQ-5D Month 3 | 3 months
  EuroQol-5D (EQ-5D) : health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated from 0 to 5 and a single summary index is obtained by summing all the dimensions (min=0 to max=25).
Quality of life Month SF-36 Month 6 | 6 months
  Quality of life assessed by the Short Form 36 version 2 (SF-36v2). The SF-36v2 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life EQ-5D Month 6 | 6 months
  EuroQol-5D (EQ-5D) : health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated from 0 to 5 and a single summary index is obtained by summing all the dimensions (min=0 to max=25).
Quality of life Month SF-36 Month 9 | 9 months
  Quality of life assessed by the Short Form 36 version 2 (SF-36v2). The SF-36v2 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life EQ-5D Month 9 | 9 months
  EuroQol-5D (EQ-5D) : health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated from 0 to 5 and a single summary index is obtained by summing all the dimensions (min=0 to max=25).
Quality of life Month SF-36 Month 12 | 12 months
  Quality of life assessed by the Short Form 36 version 2 (SF-36v2). The SF-36v2 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Quality of life EQ-5D Month 12 | 12 months
  EuroQol-5D (EQ-5D) : health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated from 0 to 5 and a single summary index is obtained by summing all the dimensions (min=0 to max=25).
Steroids Month 3 | 3 months
  Percentage of subjects with an average dose of prednisone reduced by 25% compared to M0
Steroids Month 6 | 6 months
  Percentage of subjects with an average dose of prednisone reduced by 25% compared to M0
Steroids Month 9 | 9 months
  Percentage of subjects with an average dose of prednisone reduced by 25% compared to M0
Steroids Month 12 | 12 months
  Percentage of subjects with an average dose of prednisone reduced by 25% compared to M0

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farge D, Biard L, Weil B, Girault V, Lansiaux P, Munia I, Loisel S, Charles C, Saout J, Resche-Rigon M, Korganow AS, Beuvon C, Pugnet G, Cacciatore C, Abisror N, Taupin JL, Cras A, Lowdell MW, Tarte K. Allogeneic umbilical cord-derived mesenchymal stromal cells as treatment for systemic lupus erythematosus: a single-centre, open-label, dose-escalation, phase 1 study. Lancet Rheumatol. 2025 Apr;7(4):e261-e273. doi: 10.1016/S2665-9913(24)00298-4. Epub 2024 Dec 17. PMID 39706212